CLINICAL TRIAL: NCT05453045
Title: Pharmacokinetics and Excretion of Albendazole and Its Metabolites in Saliva in Healthy Volunteers
Brief Title: Pharmacokinetics and Excretion of Albendazole and Its Metabolites in Saliva
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Nacional de Salta (Other)
Collaborators: Fundacion Mundo Sano (Unknown)
Responsible Party: Principal Investigator, Alejandro Krolewiecki, Researcher, Universidad Nacional de Salta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ABZ0301
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pharmacological Action
MeSH Terms: interventions — Albendazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Albendazole (Experimental): 400 mg po single dose
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Albendazole — tablet administration after a meal contaning approximate 15 g of fat
  Other Names: Albendazole tablet, Albendazole 400mg po

SUMMARY:
This project will develop and assess the feasibility and acceptability of a salive-based assay to monitor adherence to Mass Drug Administration (MDA) campaigns within Soil-transmitted helminthiasis (STH) control programs, evaluating the salive and serum pharmacokinetics of ALBENDAZOLE (ABZ) and its metabolites.The final goal is to obtain a field ready tool for the measurement of adherence to anthelmintic treatment at a community level that serves as a coverage/adherence indicator and a reference standard for other monitoring tools.

ELIGIBILITY:
Inclusion Criteria:

Body Mass Index: 18 to 25.

Physical exam without significant abnormal findings.

Exclusion Criteria:

Pregnancy

Lactation

Use of ABZ or other benzimidazole drugs in the previous 30 days

History of intolerance to ABZ

Malabsorption and/or other gastrointestinal conditions that might compromise ABZ absorption.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07-18 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
Salive albendazole levels | 72 hours
  Albendazole and its metabolites will be measured in salive samples through high performance liquid chromatography (HPLC).

IPD SHARING:
Plan to Share IPD: No